CLINICAL TRIAL: NCT03775772
Title: Oral Health, Bite Force and Dementia - A Randomized Controlled Clinical Trial
Brief Title: Oral Health, Bite Force and Dementia
Acronym: OrBiD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017_OrBiD_RCT
Record Dates: First submitted 2017-06-23; First posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Dementia; Oral Hygiene; Chewing Problem
Keywords: oral health; bite force; chewing efficiency; dementia; elderly; aged
MeSH Terms: conditions — Dementia | interventions — Oral Health; Bite Force

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Health - Test Group (Other): - study population is randomly assigned to control and test group
  Interventions: Procedure: Oral Health
- Bite Force/Chewing Efficacy-Test Group (Other): - study population is randomly assigned to control and test group
  Interventions: Procedure: Bite Force

INTERVENTIONS:
Procedure: Oral Health — * test group will receive an dental hygiene program for one year
  * control group will remain with dental hygiene regime like done before study participation (maximum of two dental hygiene Treatments per year)
  Arms: Oral Health - Test Group
Procedure: Bite Force — * test group will receive physiotherapy with the aim of increasing muscle strength in chewing muscles for 3 months
  * control group will remain without such training
  Arms: Bite Force/Chewing Efficacy-Test Group

SUMMARY:
Study aims: The primary aim is to identify influencing variables on oral hygiene / oral health and bite force in patients with dementia.

ELIGIBILITY:
Inclusion Criteria:

* > 59 years
* no acute processes being present
* no known cranio-mandibular dysorder (CMD) or finding of any CMD during study participation
* non or Maximum of one dental hygiene treatment in the last 12 months

Exclusion Criteria:

* younger than 60 years
* acute processes in the oral-facial Region
* known CDM case
* more than one dental hygiene treatment in the last 12 months

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Oral Health (dental examination) | 1 year
  Decayed, Missing, Filled - Index (dmf/t)
Chewing function I (examination with force gauge meter) | 1 year
  Bite Force (Bite Force Meter in Newton)

SECONDARY OUTCOMES:
Nutrition I (questionnaire/ assessment of nutritional state) | 1 year
  Mini Nutritional Assessment (MNA) (Malnutrition present? yes/no/at risk)
Nutrition II (examination for weight and body-size) | 1 year
  Body Mass Index (BMI) (normal weight / under-weight / over-weight)
Chewing function II (two-coloured chewing gum to test efficacy) | 1 year
  Chewing Efficacy (chew two-coloured chewing gum 20 times, visual and optoelectronic evaluation)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Kunze, Dr., Principal Investigator — University of Zurich
Locations (1):
- Clinic of General, Special Care and Geriatric Dentistry, Zurich, Switzerland

REFERENCES:
- [Derived] Jockusch J, Hahnel S, Nitschke I. Use of handgrip strength measurement as an alternative for assessing chewing function in people with dementia. BMC Geriatr. 2022 Sep 24;22(1):769. doi: 10.1186/s12877-022-03452-2. PMID 36153477
- [Derived] Jockusch J, Hopfenmuller W, Nitschke I. Influence of cognitive impairment and dementia on oral health and the utilization of dental services : Findings of the Oral Health, Bite force and Dementia Study (OrBiD). BMC Oral Health. 2021 Aug 14;21(1):399. doi: 10.1186/s12903-021-01753-3. PMID 34391408